CLINICAL TRIAL: NCT00211107
Title: A Placebo-Controlled, Double-Blind, Randomized, Parallel Study Of The Efficacy And Safety Of Dapoxetine HCl In The Treatment Of Rapid Ejaculation
Brief Title: A Study of the Effectiveness and Safety of Dapoxetine in the Treatment of Men With Premature Ejaculation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006088
Record Dates: First submitted 2005-09-15; First posted 2005-09-21 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Ejaculation
Keywords: dapoxetine; rapid ejaculation; premature ejaculation; ejaculation; sexual dysfunction; orgasmic disorder; sexual intercourse
MeSH Terms: conditions — Premature Ejaculation; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Coitus | interventions — dapoxetine

INTERVENTIONS:
Drug: Dapoxetine

SUMMARY:
The primary purpose of the study is to demonstrate that dapoxetine can prolong intravaginal ejaculatory latency time (IELT) compared with placebo in men with premature ejaculation (PE).

DETAILED DESCRIPTION:
One form of male sexual dysfunction is premature ejaculation (PE), which is also referred to as rapid ejaculation (RE). An objective measurement of PE in clinical studies is the intravaginal ejaculatory latency time (IELT). This is a randomized, double-blind study in men with PE. The study consists of 2 phases: pre-randomization phase (a screening visit and a 2-week baseline period); 12-week double-blind treatment phase during which patients will receive dapoxetine at one of two dosages, or placebo, for use on an "as-needed" basis. The total duration of the study is approximately 14 weeks. Patients and their partners are expected to attempt sexual intercourse at least 4 times during the baseline period and at least 6 times each month during the treatment phase. Assessments of effectiveness include the average Intravaginal Ejaculatory Latency time (IELT), as measured by stopwatch, during sexual intercourse for the treatment period (12 weeks); control over ejaculation, satisfaction with sexual intercourse, and severity of symptoms, based on questions asked at monthly intervals through the treatment phase. Safety assessments include the incidence, severity, and type of adverse events throughout treatment (12 weeks), vital sign measurements (pulse and blood pressure) and laboratory tests (hematology, chemistry, urinalysis) at monthly intervals. The study hypothesis is that treatment for 12 weeks with dapoxetine prolongs intravaginal ejaculatory latency time, compared with placebo, in men with PE. Oral tablets of dapoxetine (30 milligrams[mg] or 60mg) taken as needed during 12 weeks of treatment. No more than one dose within a 24-hour period.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual male in a stable, monogamous, sexual relationship with a female partner for at least 6 months
* onset of orgasm and ejaculation occurs with minimal sexual stimulation before or shortly after penetration and before the person wishes it
* premature ejaculation (PE) in the majority of intercourse experiences in the 6 months before study initiation
* intravaginal latency ejaculatory time (IELT) of <=2 minutes in at least 3 out of 4 events
* participants with partners of child-bearing potential must consent to use a medically acceptable method of contraception throughout the entire study
* participant's partner must have a negative pregnancy test at time of screening.

Exclusion Criteria:

* History of surgery or injury to the pelvis or spinal cord, chronic inflammation of the prostate or urethra
* taking medications that are contraindicated for participation in the study
* currently using other forms of therapy for treatment of PE (for example, behavioral therapy or medications applied locally)
* previously participated in a drug study involving dapoxetine or in another drug trial within the last month
* taken pimozide, astemizole, or monoamine oxidase inhibitors within 6 months of the start of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1294 (Actual)
Dates: Start 2003-06; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Average intravaginal ejaculatory latency time (IELT), as measured by stopwatch during sexual intercourse, between last 2 visits during the treatment period

SECONDARY OUTCOMES:
Control over ejaculation, satisfaction with sexual intercourse, and severity of symptom impressions, based on questions asked at start of study and through Week 12; incidence, severity, and type of adverse events throughout study (12 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Result] Pryor JL, Althof SE, Steidle C, Rosen RC, Hellstrom WJ, Shabsigh R, Miloslavsky M, Kell S; Dapoxetine Study Group. Efficacy and tolerability of dapoxetine in treatment of premature ejaculation: an integrated analysis of two double-blind, randomised controlled trials. Lancet. 2006 Sep 9;368(9539):929-37. doi: 10.1016/S0140-6736(06)69373-2. PMID 16962882
- [Derived] McMahon CG, Althof SE, Kaufman JM, Buvat J, Levine SB, Aquilina JW, Tesfaye F, Rothman M, Rivas DA, Porst H. Efficacy and safety of dapoxetine for the treatment of premature ejaculation: integrated analysis of results from five phase 3 trials. J Sex Med. 2011 Feb;8(2):524-39. doi: 10.1111/j.1743-6109.2010.02097.x. Epub 2010 Nov 8. PMID 21059176
- See also: A Placebo-Controlled, Double-Blind, Randomized, Parallel Study of the Efficacy and Safety of Dapoxetine HCl in the Treatment of Rapid Ejaculation — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=105&filename=CR006088_CSR.pdf